CLINICAL TRIAL: NCT04189458
Title: The Effect of a Multimodal Exercise Program on Brain Dynamics, Cognitive Functioning and Physical Fitness in Community-dwelling Older Adults
Brief Title: Multimodal Exercise Effect on Brain Dynamics, Cognitive Functioning and Physical Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Collaborators: São João de Deus School of Nursing (Unknown); Horizon 2020 - Portugal 2020 (ALT20-03-0145-FEDER-000007 - Project: ESACA) (Unknown)
Responsible Party: Principal Investigator, Hugo Filipe Zurzica Rosado, Principal Investigator, University of Évora
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Brain Dynamics
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Community-dwelling Older Adults
Keywords: Older adults; Multimodal exercise program; Brain dynamics; Cognitive functioning; Physical fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal exercise program (Experimental): The experimental group intervention will attend the multimodal exercise program. The program integrates 3 sessions / week of 60 minutes on alternated days. The multimodal exercise program includes exercises promoting simultaneous motor and cognitive stimulation.
  Interventions: Other: Multimodal exercise program
- Control Group (No Intervention): Usual care. After the study, it will be offered the opportunity to integrate a similar exercise program for the control group (CG) participants.

INTERVENTIONS:
Other: Multimodal exercise program — Each session includes: beginning ritual (5 min), warm-up (15 min), main section comprising the multimodal exercises (30 min), cool-down (5 min), and finishing ritual (5 min). At the initial stage, the activation of different muscle groups will be performed. The main section (multimodal exercises) will be focused on the specific objectives through sensorimotor and neurocognitive activities and will privilege IPS. This section includes periods ranging 10-15 min of exercises mainly focused on motor stimulation - physical fitness (strength, balance and agility) - alternating with exercises mainly focused on cognitive stimulation - CF (planning ability, solving-problems, IPS, attention and DT performance). At the cool-down the participants will normalize their physiological parameters. Finally, at the finishing ritual the participants sign an attendance sheet regarding the session, including perceived exertion (Borg Scale) and satisfaction (Caregiver Treatment Satisfaction questionnaire).
  Arms: Multimodal exercise program

SUMMARY:
The aim of present study is to analyze the effect of a multimodal exercise program on brain dynamics, cognitive functioning and physical fitness in community-dwelling older adults This experimental study is a controlled trial. Participants will be allocated to two groups: experimental group (who attend the multimodal exercise program) and control group (who maintain usual activity).

The multimodal exercise program will run for 12 weeks (3 sessions / week of 60 minutes).

Participants will be assessed 1) at baseline and at 2) at 12 weeks.

DETAILED DESCRIPTION:
Aging is associated with a decline in cognitive functioning (CF), which influence negatively the motor capacities of older adults (1). Differences on dynamic brain, namely reductions in structural and functional connectivity contribute to cognitive decline. However, efficient communications between brain regions works like a prerequisite for CF (2,3).

Programs targeting cognitive functioning improvement evidenced the importance of the information processing speed (IPS). However, IPS may not be the only factor conditioning the relationship between CF and gait in the older people, especially in locomotive tasks that require attention (4). According to Lezak et al. (5), the performance in each area of CF decreases with aging, and the most significant decline is reported on the performance of complex attentional tasks such as selective or divided attention.

Recent studies focusing cognitive or physical fitness programs, have been shown that dual-task (DT) performance, particularly involving walking while performing a task with cognitive interference, predicts the risk of frailty, disability and mortality in older people (6,7).

According Bahureksa, et al. (8), for balance maintenance is needed to incorporate and decipher the sensorimotor information through CF. On the other hand, exercise programs reported as effective strategies for agility, muscle strength and body composition improvement (9, 10). However, no studies were found focusing the effect and benefits of a multimodal exercise program privileging IPS on brain electrical activity, CF and functional fitness in community-dwelling older adults.

This multimodal exercise program, privileging information processing speed and comprising sensorimotor and neurocognitive exercises, may revert the process of loss and decline on brain dynamics, CF and physical fitness in community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥65 years;
* Community-dwelling older adults living independently;

Exclusion Criteria:

* Presence of cognitive impairment (Mini-Mental State Examination) (11);
* Presence of motor impairment compromising the program participation;
* Presence of neurological problems or diseases compromising the program participation;

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline, between and within groups comparison | 0, 3 months
  Dynamic Brain Outcome Measure - Electroencephalographic evaluation to assess frequency analyses in the alpha, theta and beta power spectrum
Change from Baseline, between and within groups comparison | 0, 3 months
  Cognitive Functioning Outcome Measure - Tower of London test, ranging from 0 (worst) to 36 (best), to assess problem-solving ability (n)
Change from Baseline, between and within groups comparison | 0, 3 months
  Cognitive Functioning Outcome Measure - Tower of London test to assess planning and execution time (s)
Change from Baseline, between and within groups comparison | 0, 3 months
  Cognitive Functioning Outcome Measure - Useful Field of View Assessment, ranging from 17 (best) to 500 (worst), to evaluate processing speed, selective and divided attention (ms)
Change from Baseline, between and within groups comparison | 0, 3 months
  Physical Fitness Outcome Measure - Timed Up and Go test (single and dual-task version) to assess agility and dual-task performance (s)
Change from Baseline, between and within groups comparison | 0, 3 months
  Physical Fitness Outcome Measure - The Ten Step Test to assess agility (s)
Change from Baseline, between and within groups comparison | 0, 3 months
  Physical Fitness Outcome Measure - Senior Fitness Test (30-Second Chair Stand) to assess lower body strength (resistance) (n)
Change from Baseline, between and within groups comparison | 0, 3 months
  Physical Fitness Outcome Measure - Short Physical Performance Battery (Chair Stand Test) to assess lower body strength (power) (n)
Change from Baseline, between and within groups comparison | 0, 3 months
  Physical Fitness Outcome Measure - Fullerton Advanced Balance Scale (modified version), ranging from 0 (worst) to 16 (best) points, to assess balance
Change from Baseline, between and within groups comparison | 0, 3 months
  Body Composition Outcome Measure - Bioimpedance analyzer (Tanita® MC-780) to assess body fat mass (%)
Change from Baseline, between and within groups comparison | 0, 3 months
  Body Composition Outcome Measure - Bioimpedance analyzer (Tanita® MC-780) to assess body lean mass (%)
Change from Baseline, between and within groups comparison | 0, 3 months
  Body Composition Outcome Measure - Bioimpedance analyzer (Tanita® MC-780) to assess body water (%)

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Rosado, MSc, Principal Investigator — University of Évora
Locations (1):
- Universidade de Évora, Evora, Portugal

REFERENCES:
- [Background] Lezak MD, Howieson DB, Bigler ED, Tranel, D. Neuropsychological assessment. New York: Oxford University Press, 5th Edition; 2012.
- [Background] Morgado J, Rocha CS, Maruta C, Guerreiro M, Martins, IP. New normative values of Mini-mental State Examination. Sinapse: Sociedade Portuguesa de Neurologia. 2009 Nov; 9(2): 10-16
- [Result] Bherer L. Cognitive plasticity in older adults: effects of cognitive training and physical exercise. Ann N Y Acad Sci. 2015 Mar;1337:1-6. doi: 10.1111/nyas.12682. PMID 25773610
- [Result] Ferreira LK, Busatto GF. Resting-state functional connectivity in normal brain aging. Neurosci Biobehav Rev. 2013 Mar;37(3):384-400. doi: 10.1016/j.neubiorev.2013.01.017. Epub 2013 Jan 17. PMID 23333262
- [Result] Bennett IJ, Madden DJ. Disconnected aging: cerebral white matter integrity and age-related differences in cognition. Neuroscience. 2014 Sep 12;276:187-205. doi: 10.1016/j.neuroscience.2013.11.026. Epub 2013 Nov 23. PMID 24280637
- [Result] Holtzer R, Mahoney J, Verghese J. Intraindividual variability in executive functions but not speed of processing or conflict resolution predicts performance differences in gait speed in older adults. J Gerontol A Biol Sci Med Sci. 2014 Aug;69(8):980-6. doi: 10.1093/gerona/glt180. Epub 2013 Nov 27. PMID 24285744
- [Result] Verghese J, Holtzer R, Lipton RB, Wang C. Mobility stress test approach to predicting frailty, disability, and mortality in high-functioning older adults. J Am Geriatr Soc. 2012 Oct;60(10):1901-5. doi: 10.1111/j.1532-5415.2012.04145.x. Epub 2012 Sep 24. PMID 23002714
- [Result] Brustio PR, Magistro D, Zecca M, Rabaglietti E, Liubicich ME. Age-related decrements in dual-task performance: Comparison of different mobility and cognitive tasks. A cross sectional study. PLoS One. 2017 Jul 21;12(7):e0181698. doi: 10.1371/journal.pone.0181698. eCollection 2017. PMID 28732080
- [Result] Bahureksa L, Najafi B, Saleh A, Sabbagh M, Coon D, Mohler MJ, Schwenk M. The Impact of Mild Cognitive Impairment on Gait and Balance: A Systematic Review and Meta-Analysis of Studies Using Instrumented Assessment. Gerontology. 2017;63(1):67-83. doi: 10.1159/000445831. Epub 2016 May 13. PMID 27172932
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Latorre Roman PA, Garcia-Pinillos F, Huertas Herrador JA, Cozar Barba M, Munoz Jimenez M. Relationship between sex, body composition, gait speed and body satisfaction in elderly people. Nutr Hosp. 2014 Oct 1;30(4):851-7. doi: 10.3305/nh.2014.30.4.7669. PMID 25335673